CLINICAL TRIAL: NCT02663011
Title: Language Error Type Evaluation in Developmental Delay Preschool Children by PLS-C
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N201508007
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Language Error Type

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- 5YR boy
  Interventions: Other: Language Evaluation-Preschool Language Scale Corrected edition(PLS-C), Lin
- 5YR girl
  Interventions: Other: Language Evaluation-Preschool Language Scale Corrected edition(PLS-C), Lin
- 4YR boy
  Interventions: Other: Language Evaluation-Preschool Language Scale Corrected edition(PLS-C), Lin
- 4YR girl
  Interventions: Other: Language Evaluation-Preschool Language Scale Corrected edition(PLS-C), Lin
- 3YR boy
  Interventions: Other: Language Evaluation-Preschool Language Scale Corrected edition(PLS-C), Lin

INTERVENTIONS:
Other: Language Evaluation-Preschool Language Scale Corrected edition(PLS-C), Lin — To assess age and gender effect in the language error type (semantics, syntax and pragmatics)of developmental delay preschool aged children, a standardize tool "Preschool Language Scale Corrected edition(PLS-C), Lin" was adopted for evaluation.

SUMMARY:
Purpose:

To assess age and gender effect in the language error type (semantics, syntax and pragmatics)of developmental delay preschool aged children, a standardize tool "Preschool Language Scale Corrected edition(PLS-C), Lin" was adopted for evaluation.

Methods:

This is a retrospective chart study enrolled 55 children aged 3, 4 and 5 in department of rehabilitation in Taipei Medical University Hospital from 2011 Jan to 2014 Dec whose average PLS-C score was at least 1.5 SD below normal. Those normal or PLS-C score was less than 1.5SD below normal were excluded. We recorded correct percentage in pragmatics, syntax, and semantics in different age group separately in auditory comprehension, language expression as well as overall performance. All wrong questions answered in PLS-C were recorded. We used SAS 9.4 (Anova, t-test) to analyze the results in age differences, gender differences, and language components differences

Results:

In overall performance, expression, and comprehension, there was no difference between boy and girl by t-test in all ages. By one-way Anova Bonferroni t test, age 5 was better than age 4 and age 3 significantly in pragmatics, syntax and semantics (p<0.005).

We further separated into groups of 5YR boy, 5YR girl, 4YR boy, 4YR girl, and 3YR boy.

In overall performance, by Duncan's multiple analysis, only 5 YR boy had significant better performance than 4 YR girl and 3 YR boy in pragmatics. In age 5, boys had better performance in pragmatics than girls (p<0.05). In age 4, no differences are showed between boy and girl.

In comprehension, in age 5, boys have better performance in pragmatics than girls(p<0.05).

In expression, there was no difference between boys and girls. Pragmatics was better than syntax (p=0.0202<o.o5) in age 5.

Conclusion:

We found age had more effect than gender in language delay children. Age 5 boys had better performance in pragmatics conflicted with some previous studies and may need more exploration in the future.

Key words:

Development Delay, Preschool aged children, Language Development Delay, Semantics, Syntax, Pragmatics, Language error type

DETAILED DESCRIPTION:
Purpose:

To assess age and gender effect in the language error type (semantics, syntax and pragmatics)of developmental delay preschool aged children, a standardize tool "Preschool Language Scale Corrected edition(PLS-C), Lin" was adopted for evaluation.

Methods:

This is a retrospective chart study enrolled 55 children aged 3, 4 and 5 in department of rehabilitation in Taipei Medical University Hospital from 2011 Jan to 2014 Dec whose average PLS-C score was at least 1.5 SD below normal. Those normal or PLS-C score was less than 1.5SD below normal were excluded. We recorded correct percentage in pragmatics, syntax, and semantics in different age group separately in auditory comprehension, language expression as well as overall performance. All wrong questions answered in PLS-C were recorded. We used SAS 9.4 (Anova, t-test) to analyze the results in age differences, gender differences, and language components differences

Results:

In overall performance, expression, and comprehension, there was no difference between boy and girl by t-test in all ages. By one-way Anova Bonferroni t test, age 5 was better than age 4 and age 3 significantly in pragmatics, syntax and semantics (p<0.005).

We further separated into groups of 5YR boy, 5YR girl, 4YR boy, 4YR girl, and 3YR boy.

In overall performance, by Duncan's multiple analysis, only 5 YR boy had significant better performance than 4 YR girl and 3 YR boy in pragmatics. In age 5, boys had better performance in pragmatics than girls (p<0.05). In age 4, no differences are showed between boy and girl.

In comprehension, in age 5, boys have better performance in pragmatics than girls(p<0.05).

In expression, there was no difference between boys and girls. Pragmatics was better than syntax (p=0.0202<o.o5) in age 5.

Conclusion:

We found age had more effect than gender in language delay children. Age 5 boys had better performance in pragmatics conflicted with some previous studies and may need more exploration in the future.

Key words:

Development Delay, Preschool aged children, Language Development Delay, Semantics, Syntax, Pragmatics, Language error type

ELIGIBILITY:
Inclusion Criteria:

* Enrolled 55 children aged 3, 4 and 5 in department of rehabilitation in Taipei Medical University Hospital from 2011 Jan to 2014 Dec whose average PLS-C score was at least 1.5 SD below normal.

Exclusion Criteria:

* Those normal or PLS-C score was less than 1.5SD below normal were excluded.

Ages: 3 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a retrospective chart study enrolled 55 children aged 3, 4 and 5 in department of rehabilitation in Taipei Medical University Hospital from 2011 Jan to 2014 Dec whose average PLS-C score was at least 1.5 SD below normal. Those normal or PLS-C score was less than 1.5SD below normal were excluded.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
What's the difference of language error types between boy and girl. | 2011 Jan to 2014 Dec
  In overall performance, expression, and comprehension, there was no difference between boy and girl by t-test in all ages.